CLINICAL TRIAL: NCT05836532
Title: Long Term Results of Surgical and Percutaneous Double Orefices Mitral Repair in Patient With p2 Prolapse Causing Degenerative Mitral Regurgitation
Status: Completed | Type: Observational
Sponsor: Michele De Bonis (Other)
Responsible Party: Sponsor-Investigator, Michele De Bonis, Chief od Cardiac Surgery of Advanced and Research Therapies, Ospedale San Raffaele
Organization: Ospedale San Raffaele (Other)
Other Study IDs: LORD-P2_DMR
Record Dates: First submitted 2023-01-26; First posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Degenerative Mitral Valve Disease; Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Central edge-to-edge — Suture of free margins of the mitral leaflets in central position to restore coaptation

SUMMARY:
Mitral regurgitation is a pathology affecting the left atrioventricular valve that causes a volumetric and pressure overload in the left chambers due to the loss of unidirectionality normally guaranteed by the cardiac valve system. The gold standard for severe mitral regurgitation is currently mitral valve plastic surgery.

Edge to edge, on the other hand, allows shorter CEC and aortic clamping times and does not require significant surgical experience in the field of mitral valve repair, therefore edge to edge could be an excellent strategy in patients suffering from mitral regurgitation caused by P2 prolapse when quadrangular resection cannot be performed.

The main objective of the present study is to examine the medium to long-term outcomes (in terms of survival and plastic outcomes) of patients undergoing central edge-to-edge to treat posterior flap pathology (P2).

ELIGIBILITY:
Inclusion Criteria:

* Mitral regurgitation with degenerative etiology
* Mitral pathology exclusively dependent on P2
* Surgical creation of a double mitral valve orifice with or without a ring as the only mitral valve repair technique.

Exclusion Criteria:

- Other mitral regurgitation etiologies (eg. functional, radiation-induced, rheumatic...)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with degenerative MR, due to P2 prolapse, who underwent surgery with central edge to edge
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2019-10-05 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
MR 2+ or more recurrency | through study completion, a minimum of 2 years

SECONDARY OUTCOMES:
Reintervention | through study completion, a minimum of 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele - Cardiac Surgery Department, Milan, Italy

IPD SHARING:
Plan to Share IPD: No